CLINICAL TRIAL: NCT06003816
Title: Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7) Water, Sanitation, and Hygiene (WASH) Case Area Targeted Intervention (CATI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Research Training and Management International (RTMI) (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00009931; 1R01AI148332-01 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Cholera; Diarrhea
Keywords: randomized controlled trial; water; sanitation; hygiene; case area targeted intervention; Bangladesh
MeSH Terms: conditions — Cholera; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7) CATI (Experimental): The CHoBI7 program is first delivered during group sessions by a health promoter to those residing in a ring around a cholera patient. The health promoter delivers a pictorial WASH module on how diarrhea can spread, and instructions on handwashing with soap, water treatment, and safe water storage. A cholera prevention package is provided containing: a one-month supply of chlorine tablets for water treatment, a soapy water bottle for handwashing, a handwashing station, and a water vessel with a lid and tap to ensure safe water storage. After the group session, households receive weekly voice and text messages from the CHoBI7 mHealth program over 12 months on the recommended WASH behaviors.
  Interventions: Behavioral: Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7) CATI
- Standard Message Arm (Active Comparator): Standard message given in the Bangladesh to diarrhea patients at health facility discharge on use of oral rehydration solution
  Interventions: Behavioral: Standard message

INTERVENTIONS:
Behavioral: Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7) CATI — The CHoBI7 program is during group sessions by a health promoter to those residing in a ring around a cholera patient reinforced through weekly voice and text messages from the CHoBI7 mHealth program over 12 months on the recommended water, sanitation, and hygiene behaviors.
  Arms: Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7) CATI
Behavioral: Standard message — Standard message given in the Democratic Republic of the Congo to diarrhea patients at health facility discharge on use of oral rehydration solution
  Arms: Standard Message Arm

SUMMARY:
Objective: The investigators objective is to develop and evaluate the effectiveness of a case area targeted water, sanitation, and hygiene (WASH) intervention in reducing cholera infections and increasing sustained WASH behaviors in transmission hotspots in a ring around cholera cases.

DETAILED DESCRIPTION:
Background: Worldwide there are estimated to be 2.9 million cholera cases annually. Effective targeted water, sanitation, and hygiene (WASH) interventions are urgently needed to reduce cholera globally. The investigators study in Bangladesh found that individuals living within 50 meters of a cholera patient were at 30 times higher risk of developing cholera than the general population during the first week after the index patient sought care at a health facility. However, there has been little work done to develop and evaluate interventions for this high risk population.

Objective: The investigators objective is to develop and evaluate the effectiveness of a case area targeted WASH intervention in reducing cholera infections and increasing sustained WASH behaviors in transmission hotspots in a ring around cholera cases.

Previous studies: The investigators research group developed the Cholera-Hospital-Based-Intervention-for-7-Days (CHoBI7), a WASH intervention delivered to cholera patients and the participants household members in a health facility. the investigators randomized controlled trial (RCT) in Bangladesh of CHoBI7 demonstrated this intervention was effective in significantly reducing cholera, and led to sustained increases in handwashing with soap and improved drinking water quality 12 months post-intervention in cholera patient households. This intervention, however, solely focused on cholera patients households. There are no studies to date that have evaluated the impact on reducing cholera of delivering a ring WASH intervention to households living near cholera patients.

Design and Setting: The Director of Disease Control at the Bangladesh Ministry of Health and Family Welfare would like to take CHoBI7 to scale across Bangladesh, and has requested the investigators build evidence on scalable approaches for delivering CHoBI7 as a CATI in a ring around cholera patient households. This study will have 3 phases. During the formative research and planning phase the investigators will develop a scalable, theory and evidence based ring WASH intervention through in-depth interviews, focus group discussions, workshops, and a pilot. During the intervention implementation and evaluation phase the investigators will conduct a RCT to prospectively follow 3120 participants from 1040 households living in 40 rings around cholera cases to evaluate the effectiveness of the intervention in: (1) reducing cholera infections during the first week after the index patient in the ring seeks care at a health facility; and (2) increasing handwashing with soap and stored water quality over a 12 month period. The first arm will receive the standard recommendation given in Bangladesh during diarrhea outbreaks on oral rehydration solution use and a leaflet on WASH practices during a single visit. The second arm will receive this message and the ring WASH intervention which includes group sessions and home visits and mobile health messages. Whole genome sequencing will be performed on water and clinical Vibrio cholerae strains collected to investigate spatiotemporal transmission dynamics of V. cholerae in hotspots. During the dissemination and policy planning phase, the investigators will partner with the Director of Disease Control to disseminate study findings and inform cholera control policies.

Significance: This will be the first RCT of a CATI WASH program to evaluate whether this intervention approach can reduce cholera.

ELIGIBILITY:
Inclusion Criteria:

* Index cholera patient have no running water inside of their home

Exclusion Criteria:

* No one will be excluded because of age, sex, religion, or sexual preference

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3140 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of non-baseline cholera infections among individuals residing in a ring around cholera patients | 1 month
  cholera infection assessed by bacterial culture and/or vibriocidal antibody titer

SECONDARY OUTCOMES:
Diarrhea among individuals residing in a ring around cholera patients | 12 months
  Self-reported or caregiver reported diarrhea (3 or more loose stools for a 24 hour period)
Child development for children under 5 years of age as assessed by the Assessed by Extended Age and Stages Assessment Questionnaire (EASQ) | 12 Months
  Assessed by Extended Age and Stages Assessment Questionnaire (EASQ)
Rate of Handwashing with soap at stool and food related events | 12 Months
  Rate of patient household members handwashing with soap at stool and food related events
Free chlorine concentration (mg/L) in stored drinking water | 12 months
  Free chlorine concentration (mg/L) in stored drinking water
Presence of Vibrio cholerae and E. coli in stored drinking water | 12 months
  E.coli and Vibrio cholerae measured by bacterial culture
Hand washing psychosocial risk factors as assessed by Water, Sanitation, and Hygiene (WASH) questionnaire | 12 months
  Water, Sanitation, and Hygiene (WASH) psychosocial risk factor questionnaire which involves both multiple choice questions and spot checks
Height-for-age measurements among children under 2 years of age | 12 months
  Height and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Height-for-age measurements among children under 5 years of age | 12 months
  Height and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age measurements among children under 2 years of age | 12 months
  Weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age measurements among children under 5 years of age | 12 months
  Weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-height measurements among children under 2 years of age | 12 months
  Height, weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards
Weight-for-height measurements among children under 5 years of age | 12 months
  Height, weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- Bangladesh (2):
  - International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka
  - Research Training and Management International, Dhaka

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified and available to our collaborators